CLINICAL TRIAL: NCT05079581
Title: Investigation of the Effects of Pelvic Floor Exercises on Pain, Sexual Dysfunction and Quality of Life in Female Patients With Sjögren
Brief Title: Pelvic Floor Exercises in Patients With Sjögren's
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Akdeniz University (Other)
Responsible Party: Principal Investigator, Sebahat Yaprak Cetin, PT, Principal Investigators, Akdeniz University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021-086
Record Dates: First submitted 2021-10-04; First posted 2021-10-15 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Sjögren; Sjögren Syndrome
Keywords: Sjögren; Pelvic floor exercises
MeSH Terms: conditions — Sjogren's Syndrome

STUDY DESIGN:
Intervention Model Description: Intervention group will perform pelvi floor exercises at home, control group will take education session
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention group (Other): Pelvic floor exercises
  Interventions: Other: Pelvic floor exercises
- Control group (No Intervention): Education session

INTERVENTIONS:
Other: Pelvic floor exercises — The participants in the intervention group will be taught exercises involving strengthening the muscles around the pelvic floor in sitting, standing and lying positions by a physiotherapist who has been trained in women's health for 4 years and will be asked to perform them as home exercises every day for 8 weeks. The exercises are as follows:
  They will be asked to tighten the muscles around the urethra, vagina and rectum as hard as possible, upwards and inwards (from the bottom up) and hold it in this way for 8-10 seconds. It will be applied in different positions as in the table.
  Arms: Intervention group

SUMMARY:
When the literature is examined, the positive effects of pelvic floor exercises on sexual functions have been supported by studies. However, the effectiveness of pelvic floor exercises on pelvic floor problems in women with sjögren has not been examined in the literature. The aim of this study is in order to examine the effect of pelvic floor exercises on sexual function in women with primer Sjögren Syndrome (pSS), since these negativities affect both the quality of life and sexual functions in women with pSS.

This is a randomized controlled trial examining the effect of 8 weeks of home-based pelvic floor exercises on pain, sexual dysfunction and quality of life on women with sjogren's.

DETAILED DESCRIPTION:
Demographic information form, HAQ, VAS, Pelvic Pain Impact Questionnaire (PPIQ), Pelvic Floor Distress Scale-20, Female Sexual Function Inventory (FSFI), Pelvic Floor Impact Questionnaire (PFIQ-7) will be applied to female patients with Sjögren's who meet the inclusion criteria.After the initial evaluation, patients will be randomized to intervention and control groups. The intervention group will be taught home exercises including fast and slow contraction and keeping the muscles around the pelvic floor in different positions (sitting, standing, lying) and will be asked to do them every day for 8 weeks according to the determined protocol. For eight weeks, the patients will be supported by the phone by the physiotherapist and at the same time, they will be checked whether they do the exercises. The control group will be given training on pelvic floor anatomy. At the end of eight weeks, patients will be given a final evaluation and the results will be analyzed.

ELIGIBILITY:
Inclusion Criteria:

* Be woman
* Having a diagnosis of primary sjogren's
* No comorbidities other than Sjögren's syndrome
* Not having had pelvic floor surgery
* Being sexually active
* Voluntary and consent to participate in the study

Exclusion Criteria:

* Other rheumatological diseases
* Urogynecological diseases
* Sarcoidosis
* lymphoma
* Having had a non-cesarean gynecological operation
* Infection

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Only female patients will be included
Enrollment: 46 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2022-08-15 (Actual); Study Completion 2022-08-15 (Actual)

PRIMARY OUTCOMES:
Pelvic Pain Impact Questionnaire | 8 weeks
  The clinical assessment of the impact of pelvic pain on women questionnaire consists of 10 questions. The first 8 questions of the questionnaire are in the form of Likert type and are scored between 0-4. The total score is reached by adding the scores given for each item, and the last two questions are not included in the calculation.
Visual Analog Scale (VAS) | 8 weeks
  It is used to convert some values that cannot be measured numerically. Two end definitions of the parameter to be evaluated are written at the two ends of a 100 mm line, and the patient is asked to indicate where on this line their situation is appropriate by drawing a line or by placing a dot or pointing. For example, for pain, I have no pain at one end and very severe pain at the other end and the patient marks his/her current state on this line. The length of the distance from the point where there is no pain to the point marked by the patient indicates the patient's pain.
Pelvic Floor Distress Scale-20 | 8 weeks
  Scale is a 20-item symptom questionnaire used to measure the degree of discomfort caused by pelvic symptoms in women. Each item consists of 4 options (Never, Rarely, Moderately, Quite often) and is scored between 1 and 4. PFDI consists of 3 sub-dimensions: Urinary distress inventory, Colo-rectal-anal distress inventory, Pelvic organ prolapse distress inventory. The mean scores of the items in each sub-dimension are calculated and these scores are multiplied by 25 and PFDI subscale scores ranging from 0-100 are calculated. Then, the 3 subscale scores are summed to find the PFDI total score, which ranges from 0-300. A higher score indicates worse health.
Female Sexual Function Inventory | 8 weeks
  This scale consists of 19 items and is a Likert type scale that evaluates sexual dysfunction in women. The validity and reliability study of FSFI was conducted by Rosen et al. (2000). The Turkish validity and reliability analysis of the scale was performed by Öksüz and Malhan (2005). The scale consists of six separate headings: desire, arousal, lubrication, orgasm, sexual success and pain. Each title is scored 0 or between 1 and 6. The lowest score is two (2) and the highest score is thirty-six (36). A higher score means better function. If the FSFI score is >30, it is classified as good, between 23-29 as moderate, and <23 as bad.

SECONDARY OUTCOMES:
Pelvic floor impact questionnaire-7 | 8 weeks
  This scale evaluates the effects of bladder, bowel and pelvic organ symptoms on an individual's activities of daily living, social relationships and emotions. Pelvic organ prolapse impact questionnaire (POPIQ-7); urinary effects questionnaire (IIQ-7); and the colorectal-anal effect questionnaire (CRAIQ-7). Each section consists of 7 questions. The questions are scored between 0 and 3 (not at all, slightly affected, moderately affected, highly affected). When calculating the total score, the average of each scale is calculated separately, multiplied by 100 and divided by 3. The scores found are summed up. The total score ranges from 0 to 300, with a low score indicating less impact of symptoms on quality of life.
Health Assessment Questionnaire | 8 weeks
  This scale is consisting of 20 questions used to question functional disability and physical disability. A high score from the scale indicates low functionality. Each item is scored between 0-3 (0: I do it with no difficulty; 1: I do it with some difficulty; 2: I do it with great difficulty; 3: I can't do it at all). In addition, the use of assistive devices and the help requested from another person are also taken into account in the scoring. The sections that make up the scale are dressing, straightening, eating, walking, hygiene, reaching, grasping and daily tasks, and each section contains two or three items. Each section is scored separately, and a single HAQ score, which can vary between 0-3, is determined by taking the average of the scores of the 8 sections. In scoring the sections, the highest score among the items forming that section is accepted as the section score.

CONTACTS AND LOCATIONS:
Locations (1):
- Antalya Training and Research Hospital, Antalya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Data will be recorded on Statistical Package Social Sciences program and then they will share only the other researches which are included in the study.

REFERENCES:
- [Result] Bo K, Talseth T, Vinsnes A. Randomized controlled trial on the effect of pelvic floor muscle training on quality of life and sexual problems in genuine stress incontinent women. Acta Obstet Gynecol Scand. 2000 Jul;79(7):598-603. PMID 10929962